CLINICAL TRIAL: NCT00446459
Title: The Highly Sensitized Patients: Effects of Mycophenolate Mofetil (MMF) On Anti-Human Leukocyte Antigen (HLA) Antibody Levels In Patients Awaiting Cadaveric Renal Transplant
Brief Title: Effects of Mycophenolate Mofetil (MMF) On Anti-HLA (Human Leukocyte Antigen)Antibody Levels In Patients Awaiting Cadaveric Renal Transplant.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. Connie Davis, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24223-A; 03-7915-A
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Kidney Failure, Chronic; Diabetic Nephropathies; Glomerulonephritis, IGA; Hypertension, Renal
Keywords: CellCept; Dialysis; Kidney; Renal; Nephropathy; Glomerulonephropathy; Immunosuppression; Allograft; Compatibility; HLA; PRA; Transplant; Sensitization; Antibodies; Diabetes; Hypertension; Transplantation, Kidney
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetic Nephropathies; Glomerulonephritis, IGA; Hypertension, Renal; Kidney Diseases; Diabetes Mellitus; Hypertension | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mycophenolate mofetil (CellCept) — 500mg - 1,000mg, taken PO, twice daily.

SUMMARY:
This is a 12-month, phase II, prospective, open label study, to evaluate the effect of mycophenolate mofetil (MMF) among patients on the kidney transplant list with high Panel of Reactive Antibody (PRA) levels.

On average, increasing the PRA from 0 to 50% specifically in the Washington Organ Procurement Organization (OPO) increases the waiting time from 3 to 6 years. Spontaneous decreases in the PRA rarely occur and is associated with a decreased chance for transplantation and a decreased rate of survival.

DETAILED DESCRIPTION:
HYPOTHESIS: mycophenolate mofetil given over 8 months to highly sensitized subjects awaiting kidney transplant, will result in a decrement in the PRA by 10% or more in approximately 40% of patients. This decrement should allow an improved rate of transplantation.

BACKGROUND: Patients who have been exposed to human tissue by prior transplants, blood transfusion or pregnancy may develop anti-bodies against the 'cell markers of human white blood cells' called 'Human Leukocyte Antigens' (HLA). Preformed anti-bodies to these foreign human tissues is called SENSITIZATION. Sensitized patients are more likely to reject a kidney from a donor who possesses the antigenic profile to which they are already sensitized. This limits the recipient's possible donor pool out of the general population.

The Panel of Reactive Antibodies (PRA) is a test panel that represents the HLA antigenic profile of the local community. The test panel is used to measure the recipient's reactivity (by percent) to a variety of HLA antigens. A PRA of 75% means the patient reacted to 75% of the antigens on the test panel. A PRA panel greater than 50% indicates that the subject (potential organ recipient) already has a significant number of antibodies pre-formed to other human tissue and is highly sensitized. Spontaneous decreases in PRA titers rarely occur thus the probability of transplantation in sensitized patients is significantly decreased.

STUDY POPULATION: adult University of Washington Medical Center patients, on the kidney transplant waiting list who are currently receiving dialysis with a PRA level over 50% and for a period of 6 months or longer.

TREATMENT PLAN/ INTERVENTION:

CONSENT: Consent will be obtained from all subjects. SCREENING: Prior to starting MMF, a thorough medical history physical exam will be obtained. Patients will be screened clinically for occurrence of infection and for protective antibodies in response to prior vaccinations and assure that they are up to date with their immunizations.

INVESTIGATIONAL PRODUCT: Mycophenolate mofetil (MMF) is used as a routine therapy for the prevention of rejection in transplant recipients and is also used routinely for the treatment of autoimmune disease and primary renal diseases such as IgA nephropathy and lupus nephritis.

HOFFMANN LA ROCHE: Will provide Mycophenolate mofetil, MMF as CellCept well as costs for laboratory testing.

DOSAGE AND ADMINISTRATION: MMF will be dispensed by investigational drug pharmacists in 250mg capsules, taken orally twice daily. Dosing of MMF will begin at 500 mg bid for 30 days then increased to 1 gm bid if subject is not experiencing undo gastrointestinal side effects or a decrease in WBC.

STUDY DESIGN:

The subjects will be continually evaluated for 12 months. Month 4: If the subject's PRA drops by 10% at month 4, subject will remain on MMF without any changes. If subject's PRA does NOT drop by 10% at month four and infections have NOT occurred, subject will remain on MMF and increase dosage if possible.

If at month four, more than 4 serious infections have occurred the MMF dose will be reduced and or stopped for that subject. If stopped they will be followed for 4 months.

Month 8:

If the subject's PRA does NOT drop by 10% at month 8, the MMF will be discontinued and the subject will be followed for the next 4 months to month 12 post enrollment.

If subject's PRA DOES drop by 10% at month 8 and NO infection(s) have occurred, subject will continue on MMF to month 12. Study subjects will be followed for a maximum of 12 months.

OBJECTIVES:

The primary endpoint:

1) The number of subjects who achieve a PRA reduction of 10% or greater within 8 months of initiating mycophenolate mofetil (MMF)therapy.

The secondary outcome measures will include:

1. The number of subjects who received a transplant during the study,
2. The number of subjects who experienced Institutional Review Board (IRB) reportable infections,
3. The number of subjects who's white blood cell count (WBC) or Immunoglobulin G or M (IgG/ IgM) titers are below range,
4. The number of transplants with a negative crossmatch.

CLINICAL AND LABORATORY EVALUATIONS:

LAB ASSESSMENT:

Immunology: PRA (panel of reactive antibodies) will be taken monthly and the levels of individual HLA anti-bodies will be evaluated every other month.

Safety:

Total levels of Immunoglobulin G (IgG) and Immunoglobulin M (IgM), as measures of the indigenous anti-body population levels. As well as HepB surface Antibody and CMV are tests done to monitor to screen for changes in the health of the subject's immune system ie. loss of memory for immunization.

A complete blood count (CBC) is taken at each visit to screen for anemia. Differential analysis on CBD for screening against platelet reduction and possible bone marrow suppression. The subject's CBC will be checked more frequently if his/her WBC, hematocrit or platelets are low. Subjects will be followed closely through 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Persons on the kidney transplant waiting list who are currently receiving hemodialysis
* Age range 18 - 75
* Outpatient status
* Patients with a PRA over 50% for over 6 months
* Patients with updated immunizations for tetanus, influenza, hepatitis B, pneumococcus
* Patients with a PPD (purified protein derivative) test within the last 6 months. If subject has a prior history of TB (tuberculosis) or positive PPD, documentation of adequate treatment is required.
* Women who are of childbearing potential must have a negative serum pregnancy test prior to being enrolled in the study and agree to use a medically acceptable method of contraception throughout the study.

Exclusion Criteria:

* Active infection
* History of multiple recurrent infections defined as more than 3 urinary tract infections, 2 episodes of pneumonia or 3 episodes of otitis/sinusitis in one year, or more than two dialysis line or peritoneal infections within one year. Infection with HCV (hepatitis C virus) or HBV (hepatitis B virus) or HIV (human immunodeficiency virus).
* Lack of documentation of PPD testing
* Lack of documentation of treatment of a positive PPD
* Pregnant or breast-feeding
* Baseline leukopenia, WBC < 4.0
* Thrombocytopenia (platelet count < 130) or difficult to treat anemia, HCT chronically < 32 on intravenous iron and EPO (erythropoietin) therapy
* Transfusion within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie L Davis, MD, Principal Investigator — University of Washington
Locations (1):
- Universtiy of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Miura S, Okazaki H, Satoh T, Amada N, Ohashi Y. Long-term follow-up of living donor renal transplant recipients sensitized after donor specific blood transfusion. Transplant Proc. 2001 Feb-Mar;33(1-2):1221-3. doi: 10.1016/s0041-1345(00)02395-2. No abstract available. PMID 11267267
- [Background] Takeda A, Uchida K, Haba T, Tominaga Y, Katayama A, Kobayashi T, Oikawa T, Morozumi K. Acute humoral rejection of kidney allografts in patients with a positive flow cytometry crossmatch (FCXM). Clin Transplant. 2000;14 Suppl 3:15-20. doi: 10.1034/j.1399-0012.2000.0140s3015.x. PMID 11092347
- [Background] Schweitzer EJ, Wilson JS, Fernandez-Vina M, Fox M, Gutierrez M, Wiland A, Hunter J, Farney A, Philosophe B, Colonna J, Jarrell BE, Bartlett ST. A high panel-reactive antibody rescue protocol for cross-match-positive live donor kidney transplants. Transplantation. 2000 Nov 27;70(10):1531-6. doi: 10.1097/00007890-200011270-00023. PMID 11118102
- [Background] Dafoe DC, Bromberg JS, Grossman RA, Tomaszewski JE, Zmijewski CM, Perloff LJ, Naji A, Asplund MW, Alfrey EJ, Sack M, et al. Renal transplantation despite a positive antiglobulin crossmatch with and without prophylactic OKT3. Transplantation. 1991 Apr;51(4):762-8. doi: 10.1097/00007890-199104000-00005. PMID 2014527
- [Background] Zanker B, Schleibner S, Schneeberger H, Krauss M, Land W. Mycophenolate mofetil in patients with acute renal failure: evidence of metabolite (MPAG) accumulation and removal by dialysis. Transpl Int. 1996;9 Suppl 1:S308-10. doi: 10.1007/978-3-662-00818-8_76. PMID 8959852
- [Background] Kaplan B, Meier-Kriesche HU, Friedman G, Mulgaonkar S, Gruber S, Korecka M, Brayman KL, Shaw LM. The effect of renal insufficiency on mycophenolic acid protein binding. J Clin Pharmacol. 1999 Jul;39(7):715-20. doi: 10.1177/00912709922008353. PMID 10392326
- [Background] Haubitz M, de Groot K. Tolerance of mycophenolate mofetil in end-stage renal disease patients with ANCA-associated vasculitis. Clin Nephrol. 2002 Jun;57(6):421-4. doi: 10.5414/cnp57421. PMID 12078944
- [Background] Gloor JM, Lager DJ, Moore SB, Pineda AA, Fidler ME, Larson TS, Grande JP, Schwab TR, Griffin MD, Prieto M, Nyberg SL, Velosa JA, Textor SC, Platt JL, Stegall MD. ABO-incompatible kidney transplantation using both A2 and non-A2 living donors. Transplantation. 2003 Apr 15;75(7):971-7. doi: 10.1097/01.TP.0000058226.39732.32. PMID 12698082
- [Background] Holechek MJ, Hiller JM, Paredes M, Rickard JC, Montgomery RA. Expanding the living organ donor pool: positive crossmatch and ABO incompatible renal transplantation. Nephrol Nurs J. 2003 Apr;30(2):195-204. PMID 12736998

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study subjects were recruited from University of Washington Medical Center's kidney transplant wait list. Patients with a Panel of Reactive Antibodies (PRA)over 50% for 6 months or longer between 18 and 75 year of age were contacted by letter and then by phone to schedule screening visit. Enrollment occured from 4/24/06 to 9/06/07.
Pre-assignment Details: Subjects were consented, given a physical exan and laboratory tests including serum virologies current Hepatitis B immunization and Tuberculosis (TB) testing initially. Abnormalities in white or red blood cells, platelets, TB test or signs of infection or evidence of cancer were grounds for exclusion.
Groups:
- Mycophenolate Mofetil (MMF) Single Arm Study: MMF mono-therapy, oral dosing of 500 - 1,000 mg twice daily as tolerated.
Period: 8 Months
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Started | 34 (34 subjects received any amount of MMF.)
Completed | 22 (22 subjects were on study at month 8.)
Not Completed | 12
Not completed — Protocol Violation | 12
Period: 12 Months
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Started | 22 (22 subjects remained on-study at month 8)
Completed | 4 (4 subjects remained at month 12)
Not Completed | 18
Not completed — Protocol Violation | 4
Not completed — 14 subjects to MMF + Rituximab Study | 14

BASELINE CHARACTERISTICS:
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Secondary Outcome: The Number of Subjects With Significant Infections up to Month 12.
Description: The number of infections while on-study up to month 12. Subjects who's PRA decreased by 10% at month 8 and who went on to the Mycophenolate mofetil + Rituximab study were followed to month 8. Those subjects who stayed on the Mycophenolate mon-therapy study were observed for infection over 12 months or until they seperated from the study.
Time Frame: From enrollment to month 12.
Population: Forty five subjects were screened, of these 37 received MMF.
Measure: Number; unit: Participants
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Participants | 4

2. Primary Outcome: The Number of Subjects With a 10% Decrease in PRA Level at Month 8.
Time Frame: Enrollment to month 8
Measure: Number; unit: Participant
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Participant | 9

3. Secondary Outcome: The Number of Kidney Transplant up to 12 Months.
Description: The number of kidney transplants up to month 12. Subjects who's PRA decreased by 10% at month 8 and who went on to the Mycophenolate mofetil + Rituximab study were followed to month 8. Those subjects who stayed on the Mycophenolate mon-therapy study were observed for infection over 12 months or until they seperated from the study.
Time Frame: Enrollment to month 8 or month 12 post enrollment.
Measure: Number; unit: Participants
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Participants | 3

4. Secondary Outcome: The Number of Pariticpants With a White Blood Cell Count Below 2.0 Thousand (Low) or Total IgG/IgM Titers Below Range (620-1490 mg/dL).
Description: The number of subjects with adverse hematologic effects with MMF while on-study. Subjects who's PRA decreased by 10% at month 8 and who went on to the Mycophenolate mofetil + Rituximab study were followed to month 8. Those subjects who stayed on the Mycophenolate mon-therapy study were observed for hematologic effects up to 12 months.
Time Frame: Enrollment to month 12.
Measure: Number; unit: Participant
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Participant | 0

5. Secondary Outcome: The Number of Transplants With a Negative Crossmatch at Transplant.
Description: The number negative crossmatch transplants up to month 12. Positivie crossmatch transplant carries a higher risk for rejection. Subjects who's PRA decreased by 10% at month 8 and who went on to the Mycophenolate mofetil + Rituximab study were followed to month 8. Those subjects who stayed on the Mycophenolate mon-therapy study were observed for negative crossmatch transplants to 12 months.
Time Frame: Number of Transplants with a Negative Crossmatch.
Measure: Number; unit: Participant
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Number analyzed (Participants) | 34
Participant | 0

ADVERSE EVENTS:
Time Frame: From enrollment to month 12.
Description: Definition of SAE: hospitalization or significant treatment or interference with ADLs.
Arm/Group | Mycophenolate Mofetil (MMF) Single Arm Study
Serious Adverse Events (participants affected / at risk) | 2/37
Other Adverse Events (participants affected / at risk) | 6/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (MMF) Single Arm Study (N=37)
Myocardial infarction (Cardiac disorders) | 1 (1) — Potasium level increase in this subject caused M.I.
Retinal stroke (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (MMF) Single Arm Study (N=37)
Peritonitis (Infections and infestations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Abscess (Infections and infestations) | 2 (3) — Abscess-folliculitis and peri-renal abscess

LIMITATIONS AND CAVEATS:
The treatment of highly sensitized patients on dialysis with single agent therapy of mycophenolate was hampered by gastrointestinal side effects that reduced anticipated maximum tolerated doses and duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days